CLINICAL TRIAL: NCT03884920
Title: Impaired Glucose Tolerance and Prevention of Diabetes Mellitus Type 2 by Polyherbal Formulation of Eastern Medicine
Brief Title: Glucose Tolerance and Prevention of Diabetes Mellitus Type 2 by Polyherbal Formulation
Acronym: Phase-1
Status: Completed | Type: Observational
Sponsor: Islamia University of Bahawalpur (Other)
Collaborators: Hashmi Herbal Pharma (HHP) Registered Bahawalpur (Unknown)
Responsible Party: Principal Investigator, Hafiz Abdul Sattar Hashmi, Principal Investigator, Islamia University of Bahawalpur
Other Study IDs: Hashmi5767
Record Dates: First submitted 2019-03-15; First posted 2019-03-21 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus; Pre Diabetes
Keywords: Impaired Fasting Glucose; Impaired Glucose Tolerance; 2hr -75gm Oral Glucose Tolerance Test; Diabetes Mellitus Prevention
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A Pre-diabetic placebo: Group of pre-diabetics receiving placebo BD for six weeks
- Group B Pre-diabetic test: Group of Pre-diabetic receiving polyherbal / test candidate 900mg in two divided doses for six weeks
  Interventions: Dietary Supplement: Polyherbal formulation
- Group C Diabetic test: Early onset of Diabetes mellitus receiving polyherbal formulation 1800mg in two divided doses for six weeks
  Interventions: Dietary Supplement: Polyherbal formulation

INTERVENTIONS:
Dietary Supplement: Polyherbal formulation — Test candidate will be administered per oral before / with meal in two divided doses
  Groups: Group B Pre-diabetic test; Group C Diabetic test

SUMMARY:
Primary protocol to this study is to develop a natural remedy to prevent diabetes mellitus in pre-diabetic state and elaborate the effectiveness of polyherbal formulation for carrying out Phase-II, III and IV. It also aimed at to see the level of difference of glucose tolerance and impaired fasting glucose and impaired glucose tolerance between pre-diabetic and diabetic to evaluate the potential benefit for treatment of insulin resistance and sensitivity. To see the for prevention of Diabetes Mellitus (DM) and stopping / delaying the onset of DM.

DETAILED DESCRIPTION:
This study is a clinical trial study to evaluate the potential of prevention in pre-diabetics and to prevent onset of diabetes mellitus. For this purpose, volunteers will be enrolled in the study by observing the Helsinki Declaration for clinical trials.

volunteers will be screened for the impaired glucose tolerance or impaired fasting glucose or at risk to develop diabetes mellitus type 2.

On screening, pre-diabetics and early onset diabetics with no previous history of treatment etc will be grouped into A and B.

Biochemical evaluations will be carried out at base line and followed by three weeks intervention and evaluation of biomarkers and at sixth week for further evaluation.

Collected data will be evaluated for primary out comes and secondary out come. statistical analysis will be done. One year followup of participants was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-59
* Impaired Fasting Glucose (100-125mg/dl)
* Impaired Glucose Tolerance (140-199mg/dl) 2h-75gm OGTT
* History of Diabetes in first degree relation with one condition
* At high risk with BMI > 35%
* Early onset diabetic / accidental on screening (glucose >200mg/dl)

Exclusion Criteria:

* on renal dialysis;
* an acute or terminal illness or serious mental illness;
* history of recent coronary event within the last 12 months;
* a recent history of acute medical problem or admission to hospital;
* any other severe medical conditions that need intervention / treatment
* has poor short-term prognosis (expected death in <2 years);
* is planning to travel for longer than 6 weeks during the 6-week intervention period; or
* is with compromised liver / kidney / cardiac function
* older patients of DM taking any form of medication / intervention

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * community samples will be obtained from the area of Bahawalpur
  * Model Town A, B, and
  * remote areas of district Bahawalpur consisting of Khairpur Tamewali city population
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Fasting Glucose Tolerance (FGT) | six weeks
  enhancement of fasting glucose tolerance (<100mg/dl)
Glucose Tolerance (GT) | six weeks
  enhancement of oral glucose tolerance (<140mg/dl)
HB-A1c | six week
  improvement in glycated hemoglobin (HB-A1c) percentage <6%,

SECONDARY OUTCOMES:
Lipid Profile | six weeks
  serum Cholesterol level (mg/dl)
Lipid Profile | Six Weeks
  Serum Triglycerides (mg/dl)
Lipid Profile | Six week
  Serum Low Density Lipids (LDL) (mg/dl)
Lipid Profile | six week
  Serum High Density Lipids (HDL) (mg/dl)

OTHER OUTCOMES:
Liver Functions | six week
  Serum Glutamate pyruvate transaminase (SGPT) (mg/dl)
Liver Function | six week
  serum glutamate oxaloacetate transaminase (SGOT)(mg/dl)
Liver Function | six week
  Alkaline phosphatase (ALP)
Kidney Function | six week
  Serum creatinine (mg/dl)
Kidney Function | six week
  Blood Urea Nitrogen (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: H A Sattar Hashmi, M.Phil, Principal Investigator — scholar; Dr K A.Ansari, Ph.D, Study Director — AP
Locations (2):
- Pakistan (2):
  - Hashmi Dawakhana, Khairpur Tamewali, Punjab Province
  - University College of Conventional Medicine, Bahawalpur

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT03884920/Prot_001.pdf